CLINICAL TRIAL: NCT00141284
Title: A Phase Iv Single-Arm Open-Label Non-Randomized Study To Evaluate The Safety And Pharmacokinetics Of Nelfinavir (Viracept, A430) 1250mg Twice Daily (250mg Or 625mg Forms) With Lamivudine/Zidovudine (Combivir) Background Therapy In Hiv/Hepatitis C Virus (Hcv) Co-Infected Subjects With Hepatic Dysfunction.
Brief Title: An Open Label Study To Evaluate The Safety and Kinetics of Nelfinavir in Subjects With HIV and Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4301003
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: HIV Infection; Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Nelfinavir; Zidovudine; Lamivudine

INTERVENTIONS:
Drug: nelfinavir 1,250 mg twice daily
Drug: Zidovudine 300 mg twice daily
Drug: Lamivudine 150 mg twice daily

SUMMARY:
The purpose of this study is to confirm the safety, efficacy and delineate the pharmacokinetic properties of nelfinavir in HIV/ Hepatitis C coinfected subjects with Child Pugh A compensated cirrhosis and or Hepatic fibrosis

ELIGIBILITY:
Inclusion Criteria:

* HIV/ Hepatitic C co infected with documented HCV viremia evidence for cirrhosis and or hepatic fibrosis on liver biopsy, positive fibrosis index, stable health

Exclusion Criteria:

* Decompensated cirrhosis (Child Pugh B or C)
* Pregnant or lactating women
* History of previous antiretrovirals > 14 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To Evaluate the safety of nelfinavir 1,250 mg orally taken twice daily in HIV/HCV co infected adult subjects with compensated cirrhosis (Child Pugh A) or hepatic fibrosis.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of nelfinavir and M8, the major metabolite.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (4):
  - Pfizer Investigational Site, Bakersfield, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Dallas, Texas
- Pfizer Investigational Site, Toronto, Ontario, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4301003&StudyName=An%20Open%20Label%20Study%20To%20Evaluate%20The%20Safety%20and%20Kinetics%20of%20Nelfinavir%20in%20%20Subjects%20with%20HIV%20and%20Hepatitis%20C%20%20%20%20